CLINICAL TRIAL: NCT06711861
Title: Multicenter Retrospective Study on Streptobacillus Moniliformis Infections in France
Acronym: Streptobacil
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9237
Record Dates: First submitted 2024-08-21; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-08

CONDITIONS: Streptobacillus Moniliformis Infections
Keywords: Streptobacillus moniliformis; Zoonosis; Rat bites; Zoonotic diseases
MeSH Terms: conditions — Rat-Bite Fever; Zoonoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
French data on Streptobacillus moniliformis infections (zoonosis transmitted by rat bites) are rare and there are no case series in the literature to date. This is a pathology presenting atypical clinical manifestations for a bacterial infection and which therefore remains underdiagnosed. Streptobacillus moniliformis infections can be fatal without appropriate antibiotic treatment. This study could improve diagnosis, develop early treatment strategies and contribute to the overall understanding of zoonotic diseases

ELIGIBILITY:
Inclusion Criteria:

* Minor patient aged 1 to 17 years
* Adult patient ≥18 years
* Proven Streptobacillus moniliformis infection between 01/01/2007 and 31/12/2023
* Subject not objecting, after being informed, to the reuse of their data for the purposes of this research
* Holders of parental authority not objecting, after being informed, to the reuse of their data for the purposes of this research their child for the purposes of this research

Exclusion Criteria:

* Subject and/or holder of parental authority having expressed opposition to participating in the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient having Streptobacillus moniliformis infection between 01/01/2007 and 31/12/2023
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-02-16 (Estimated); Study Completion 2025-02-16 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the effectiveness of antibiotic therapy initiated for the treatment of Streptobacillus moniliformis infection. | Negative blood culture 15 days after the start of antibiotic therapy.
  Clinical cure 15 days after the start of antibiotic therapy. This cure is based on a negative blood culture (absence of germs) performed 15 days after the start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France